CLINICAL TRIAL: NCT04293510
Title: Evaluation of Janus Kinase_3 Expression in Juvenile Onset Systemic Lupus Erythematosus
Brief Title: Evaluation of Janus Kinase_3 in Juvenile Onset Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, enas mohamed sayed ahmed, Principal Investigator, Assiut University
Other Study IDs: EKNL
Record Dates: First submitted 2020-02-29; First posted 2020-03-03 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Janus-kinase3; active; lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Motor Activity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — frozen renal tissue and whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group study 1: children and adolescents who diagnosed as lupus patients
  Interventions: Procedure: renal biopsy and blood sampling
- group study 2: age and sex matched healthy children free from any infection with no family history of immunological diseases

INTERVENTIONS:
Procedure: renal biopsy and blood sampling — renal biopsy and blood sampling will be taken from lupus patients for evaluation of Janus-kinase 3
  Groups: group study 1

SUMMARY:
One of the best understood mechanisms by which cytokines activate signals, thus eliciting specific responses in target cells, involves enzymes such as Janus kinases (JAKs) and transcriptional factors such as signal transducers and activators of transcription (STATs). For immune mediated diseases, both activating and inactivating mutations of JAKs and STATs may cause abnormalities in immune homeostasis. Polymorphisms of JAK/STAT genes have been linked to susceptibility for rheumatoid arthritis (RA) , systemic lupus erythematosus (SLE), psoriatic arthritis (PA) and inflammatory bowel disease (IBD) .

Janus_kinase 3 expression will be evaluated in the serum and renal tissue of lupus patients during active stage of the disease through this study

DETAILED DESCRIPTION:
Investigators will assess the relationship between the expression of Janus_kinase 3 and the clinical and laboratory parameters of disease activity . Disease activity will be assessed through the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI). Also, investigators will evaluate the relationship between Janus_ kinase 3 expression and histopathological classes of lupus nephritis according to the 2003 International Society of Nephrology/ Renal Pathology Society (ISN/RPS) classification of lupus nephritis. This will be done through Janus_kinase 3 assessment in the blood and renal tissue of lupus patients.

ELIGIBILITY:
Inclusion Criteria:

* Age younger than 16 years.

  * Active disease stage
  * Patients with biopsy proven lupus nephritis according to ISN/RPS classification criteria of lupus nephritis

Exclusion Criteria:

* Lupus patients in remission.

  * Lupus patients with end stage renal disease.
  * Lupus patients with secondary thrombotic thrombocytopenic purpura (TTP) and hemolytic uremic syndrome (HUS).
  * patients with moderate or severe infection

Ages: 7 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: This will include children and adolescents who fulfill the 2012 Systemic Lupus International Collaborating Clinics (SLICC) classification criteria of systemic lupus erythromatosus during a period of 2 years.
Sampling Method: Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Janus-kinase 3 expression | within 2 years
  evaluation of Janus-kinase 3 expression in blood and renal tissue of lupus patients during active stage of disease

SECONDARY OUTCOMES:
correlation | 2 years
  relationship between Janus- kinase expression and clinical and laboratory parameters of disease activity

OTHER OUTCOMES:
correlation | 2 years
  relationship between Janus-kinase 3 expression and histopathological classification of renal biopsy in lupus nephritis proven patients

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yamaoka K, Saharinen P, Pesu M, Holt VE 3rd, Silvennoinen O, O'Shea JJ. The Janus kinases (Jaks). Genome Biol. 2004;5(12):253. doi: 10.1186/gb-2004-5-12-253. Epub 2004 Nov 30. PMID 15575979
- [Background] Remmers EF, Plenge RM, Lee AT, Graham RR, Hom G, Behrens TW, de Bakker PI, Le JM, Lee HS, Batliwalla F, Li W, Masters SL, Booty MG, Carulli JP, Padyukov L, Alfredsson L, Klareskog L, Chen WV, Amos CI, Criswell LA, Seldin MF, Kastner DL, Gregersen PK. STAT4 and the risk of rheumatoid arthritis and systemic lupus erythematosus. N Engl J Med. 2007 Sep 6;357(10):977-86. doi: 10.1056/NEJMoa073003. PMID 17804842
- [Background] Weening JJ, D'Agati VD, Schwartz MM, Seshan SV, Alpers CE, Appel GB, Balow JE, Bruijn JA, Cook T, Ferrario F, Fogo AB, Ginzler EM, Hebert L, Hill G, Hill P, Jennette JC, Kong NC, Lesavre P, Lockshin M, Looi LM, Makino H, Moura LA, Nagata M. The classification of glomerulonephritis in systemic lupus erythematosus revisited. J Am Soc Nephrol. 2004 Feb;15(2):241-50. doi: 10.1097/01.asn.0000108969.21691.5d. PMID 14747370
- [Background] Petri M. Review of classification criteria for systemic lupus erythematosus. Rheum Dis Clin North Am. 2005 May;31(2):245-54, vi. doi: 10.1016/j.rdc.2005.01.009. PMID 15922144